CLINICAL TRIAL: NCT04309279
Title: The Effects of Zentangle on Psychological Well-being Among Adults in Hong Kong: A Pilot Randomized Controlled Trial
Brief Title: Zentangle on Psychological Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PSY011
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Mental Health Wellness
Keywords: Zentangle; Mindful doodling; Mindfulness; Psychological Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The randomization will be performed by an independent assessor using a computer-generated list of numbers. A 2-hour online Zentangle class will be delivered to the Zentangle group by a certified Zentangle teacher via online webinar. The Zentangle group will complete a short qualitative questionnaire and participate in a 15-minute brief discussion right after the Zentangle class. They will also be encouraged to practice Zentangle daily for two weeks. Both Zentangle group and waitlist control group will complete a set of online questionnaires before the intervention commences, immediately after the intervention and 2 weeks after the intervention. An online Zentangle class will be provided to the waitlist control group after the post-intervention data of the Zentangle group has been collected.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zentangle group (Experimental)
  Interventions: Behavioral: Zentangle
- Wait-list Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Zentangle — Zentangle is a mindful doodling process in which participants draw repetitive, structured patterns on small pieces of paper. The patterns consist of combinations of dots, lines, and curves.
  Other Names: Mindful doodling
  Arms: Zentangle group

SUMMARY:
This study will examine the effects of Zentangle as an intervention for reducing stress and enhancing psychological wellbeing among Hong Kong adults. Zentangle is a mindful doodling process in which participants draw repetitive, structured patterns on small pieces of paper. The patterns consist of combinations of dots, lines, and curves. Zentangle is developed in 2003 by two Americans, and this concept is still new to many people. Some studies suggested that Zentangle can be effective in reducing stress and anxiety, but the number of research papers on Zentangle is limited. Although Zentangle has become a rather popular stress relief activity in Hong Kong recently due to its easiness to learn and minimal tool requirement, there is no related study on its effectiveness in promoting psychological wellbeing in Hong Kong.

DETAILED DESCRIPTION:
This study will be a pilot randomized controlled trial on the effects of Zentangle as an intervention for reducing stress and enhancing psychological wellbeing among Hong Kong adults. Prior to all study procedures, an online informed consent (with phone support) will be obtained from potential participants. Around 30 eligible participants will be randomly assigned to either the Zentangle group or the waitlist control group in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents
2. Aged from 18 to 65
3. Cantonese language fluency
4. Willingness to provide informed consent and comply with the trial protocol
5. Be able to join online webinar via a computer

Exclusion Criteria:

1. Have suicidal ideation
2. Are using medication or psychotherapy for any psychiatric disorder
3. Experiencing depression and anxiety
4. Have major psychiatric, medical or neurocognitive disorders that make participation infeasible based on the research team's judgment
5. Are currently participating in a mindfulness practice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS) | Baseline (Pre-intervention), immediately after intervention and 2-week post-intervention
  PANAS is a 20-item scale, comprises of two 10-item subscales measuring positive affect (PA) and negative affect (NA). This self-report measure is being widely used in both clinical and community settings. A 5-point Likert scale is employed, ranging from "very slightly or not at all" to "extremely", to measure the extent to which participants have experienced such feelings over a specific period of time.

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scales-21 (DASS-21) | Baseline (Pre-intervention) and 2-week post-intervention
  DASS-21 is a 21-items scale, comprises of three sub-scales which measures the negative emotional states of depression, anxiety, and stress. The DASS is based on a dimensional rather than a categorical conception of psychological disorder; thus, it has no direct implications for the allocation of patients to discrete diagnostic categories. However, recommended cutoff scores for conventional severity labels (normal, moderate, severe) are given in the DASS Manual.
Five Facet Mindfulness Questionnaire-Short Form (FFMQ-SF) | Baseline (Pre-intervention) and 2-week post-intervention
  The FFMQ-SF is a 24-item scale that is used to evaluate one's dispositional tendency to be mindful in daily life. Ratings on the 5-point Likert scale are obtained on 5 factors, including acting with awareness, describing, nonjudging, nonreactivity and observing. The 5-point scale ranging from "never or rarely true" to "very often or always true" is used to rate how frequent the participants had each experience.
Self-Compassion Scale-Short Form (SCS-SF) | Baseline (Pre-intervention) and 2-week post-intervention
  SCS-SF is a 12-item scale to evaluates the degree of self-compassion. Ratings on the 5-point Likert scale are obtained on 6 factors, including self-kindness, common humanity, mindfulness, selfjudgment, isolation and over-identification. The self-report 12-item SCS-SF explicitly represents the thoughts, emotions, and behaviors associated with self-compassion and includes items that measure how often people respond to feelings of inadequacy or suffering with each of six components.
Insomnia Severity Index (ISI) | Baseline (Pre-intervention) and 2-week post-intervention
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Treatment evaluation form and engagement questionnaire | Immediately after intervention and 2-week post-intervention
  Treatment evaluation form and engagement questionnaire will be used to collect participants' view on the Zentangle class and how often they practiced Zentangle for the past 2 weeks respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong